CLINICAL TRIAL: NCT05385172
Title: Evaluation of the Effectiveness of the Video Prepared to Raise Cervical Cancer Awareness in Women Between the Ages of 18 and 65 Via Social Media.
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ebru Şen, PhD Student-Lecturer, Istanbul University - Cerrahpasa
Other Study IDs: E-57840365-044-1607
Record Dates: First submitted 2022-04-28; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Being a Woman Aged 18-65
Keywords: Cervical Cancer; Social Media; Awareness; HPV; Pap-smear
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 18-65 years old women
  Interventions: Other: No any intervation.

INTERVENTIONS:
Other: No any intervation. — This research, a quasi-experimental study based on the comparison of the pre-test and post-test results of individuals in a single group is conducted to raise awareness about cervical cancer in women aged 18-65 years.
  Other Names: This research, a quasi-experimental study based on the comparison of the pre-test and post-test results.

SUMMARY:
This research, a quasi-experimental study based on the comparison of the pre-test and post-test results of individuals in a single group is conducted to raise awareness about cervical cancer in women aged 18-65 years. The questionnaire includes 32 questions about the individual's socio-demographic characteristics, pregnancy, and sexual life information, cervical cancer, pap-smear test, and HPV vaccine information, as well as a 27-item 3-point likert type to measure cervical cancer risk factors, symptoms, and prevention. A survey form consisting of 61 questions, consisting of 2 questions and 2 guestions for evaluating the animated training video, and an informative animated training video of 4 minutes and 33 seconds constituted the data collection tools. During the Covid-19 pandemic, the study has completed with 433 people who participated voluntarily by directing the participants via online platforms (WhatsApp / Instagram / E-mail) using the snowball sampling method of survey applications. The women who participated in the research completed the first part by watching the informative animated training video at the end of the questionnaire form.

ELIGIBILITY:
Inclusion Criteria:

* be 18-65 years old
* Being literate
* Using Whatsapp / Instagram / Email
* Will volunteer to participate in the research.

Exclusion Criteria:

* Attending the pre-test but not participating in the post-test
* Filling the survey form incompletely.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of the study consists of women aged 18-65 living in our country. In 2018 TUIK data, it was stated that the average number of women between the ages of 18-65 was 33 million, and the minimum number of women to be reached was found to be 385, as a result of calculating the sample with a known sample, taking into account the 5% margin of error and 95% confidence level. During the Covid-19 pandemic, survey applications were directed through the online platform (WhatsApp / Instagram / E-mail) using the snowball sampling method, and 433 people who agreed to participate voluntarily between 01 April and 01 June 2021 and met the inclusion criteria constituted the sample of the research.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
Awareness level measurement about cervical cancer. | Through study completion, an average of 1 year.
  The knowledge level was measured by pre-test and post-test by watching the informative animated video prepared for the participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University - Cerrahpasa, Avcılar, Turkey (Türkiye)